CLINICAL TRIAL: NCT04431752
Title: Development of Spin-lock and FSE Acquisitions Based 3D Quantitative Biochemical Imaging for Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: 2020.115
Record Dates: First submitted 2020-05-14; First posted 2020-06-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy Volunteer: 10 healthy volunteers to undergo radiographic examinations of the knee joint.
  Interventions: Radiation: Magnetic Resonance Imaging Scan
- Kellgren-Laurence grading I Osteoarthritis Knee: 10 patients in Kellgren-Laurence grading I to undergo radiographic examinations of the knee joint.
  Interventions: Radiation: Magnetic Resonance Imaging Scan
- Kellgren-Laurence grading II Osteoarthritis Knee: 10 patients in Kellgren-Laurence grading II to undergo radiographic examinations of the knee joint.
  Interventions: Radiation: Magnetic Resonance Imaging Scan
- Kellgren-Laurence grading III Osteoarthritis Knee: 10 patients in Kellgren-Laurence grading III to undergo radiographic examinations of the knee joint.
  Interventions: Radiation: Magnetic Resonance Imaging Scan
- Kellgren-Laurence grading IV Osteoarthritis Knee: 10 patients in Kellgren-Laurence grading IV to undergo radiographic examinations of the knee joint.
  Interventions: Radiation: Magnetic Resonance Imaging Scan

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging Scan — The selection of patients with different level of OA will be made using the existing Kellgren-Laurence grading systems. The recruited patients will receive MRI exams with our enhanced sequencing. The OA level of each patient will be determined objectively through our quantitative OA grading system on MRI, which will be compared to Kellgren-Laurence grading results to evaluate the clinical performance of the MRI.

SUMMARY:
In Hong Kong, joint diseases are common health problems as identified by the Elderly Health Service under the Department of Health. It accounts for most of the disability of the elderly in Hong Kong. In particular, osteoarthritis (OA) is on the rise and the prevalence of OA increases with age. Women are more likely to have OA in knee and hip joints after menopause. A study in 2000 reported that among Hong Kong people aged 50 and above, 7 percent of men and 13 percent of women suffered from OA. With an ageing population, it is expected that OA will become a major public health problem in Hong Kong and worldwide and the socio-economic cost of supportive care to these patients can become a major burden to Hong Kong society and many regions in the world. Early diagnosis and prevention of OA and effective technology for treatment monitoring are very important. At present, the management of OA is not optimal and standard quality indicators suggest that the majority of persons with the disease do not receive appropriate care. Over half of the population affected with OA are unaware of the diagnosis. The research team have developed a quantitative and fully automated non-contrast MRI application for early detection and monitoring of joint diseases. The whole project was funded by the Innovation and Technology Fund (ITF) (MRP/001/18X ) started in January 2019. This clinical trial is part of the quantitative assessment of this developed technology. The team anticipate this innovation will address both OA diagnosis, surveillance and management. This can potentially increase diagnostic capabilities with minimum efforts, improving patient awareness, and improved treatment monitoring of the disease state after the interventions. Thus, the proposed technology is expected to provide betterment in the quality of life for the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* All Patients over the age of 18
* All patients must provide their written consent

In the OA group

* Patients must be affected by primary osteoarthritis of the knee (according to ACR - American College of Rheumatology - classification)
* All patients must have pain symptoms for more than or equal to 2 months
* Radiological evidence of osteoarthritis

Exclusion Criteria:

* Contraindication to MRI
* Patient with a mental disability
* Claustrophobia
* Inflammatory arthritis
* Ongoing Pregnancy and breast-feeding
* Presence of severe diseases like terminal cancers
* Presence of metalwork in the knee
* Significant hematological diseases;
* Non-consenting patients who have not provided the written Informed Consent
* Gross lower limb deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteer and Knee Osteoarthritis Patient groups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of cartilage wear | Through study completion, an average of 1 year
  All patient will have Xrays and MRI to quantitative assess the degree of cartilage wear.
  The patient will be categorised based on their Kellgren-Lawrence grading.

SECONDARY OUTCOMES:
Oxford Knee Score | Through study completion, an average of 1 year
  Clinical Questionnaire Assessment Tool. Subjective patient-reported outcome measurement (Oxford Knee Score) will be performed at the time of recruitment and prior to the MRI. Score 80-100 = Excellent, Score 70-79 = Good, Score 60-69 = Fair, Score below 60 = Poor.
Knee Society Function Score | Through study completion, an average of 1 year
  Clinical Questionnaire Assessment Tool. Score from 100 to -20. The higher the score, the better the knee function outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided